CLINICAL TRIAL: NCT04456907
Title: Systemic Effects After Local Injection of Platelet-rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6501714
Record Dates: First submitted 2020-06-02; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2017-03

CONDITIONS: Platelet Rich Plasma (PRP)
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPR group (Experimental): Receive PRP injection
  Interventions: Other: platelet rich plasma
- Saline group (Sham Comparator): Receive saline injection
  Interventions: Other: saline injection

INTERVENTIONS:
Other: platelet rich plasma — Autologous platelet-rich plasma (PRP) was prepared using the RegenKit THT system (RegenLab SA, Le Mont-sur-Lausanne, Switzerland) following the manufacturer's instructions. Medical technicians, who had been well-trained by the manufacturer, were responsible for the process of PRP preparation. For each patient, 8-10 mL of venous blood was drawn and collected to the commercial RegnLab THT tube, which contained 1 mL sodium citrate. After single centrifugation at 3400 revolutions per minute (rpm) for 8 minutes, 4-5 mL of PRP was yielded with leukocytes maintained at physiological levels and red blood cells depleted. Then, the blood components were separated, with the platelet pellet resting on the separating gel. PRP for later application was obtained by re-suspending the platelet pellet in the plasma supernatant by gently inverting the unopened RegenKit THT tube 5 to 10 times.
  Arms: PPR group
Other: saline injection — saline injection
  Arms: Saline group

SUMMARY:
Objective Platelet-rich plasma (PRP) is widely utilized in the treatment of sports injuries with favorable outcomes. However, potential systemic effects after localized PRP injection are unclear at present.

Design: prospective randomized study Methods Twenty-four Taiwanese male athletes with tendinopathy were randomized into a PRP group (n = 13) or a saline group (n = 11).

ELIGIBILITY:
Inclusion Criteria

- Adult male athletes were diagnosed with tendinitis

Exclusion Criteria:

* Receive local injections and surgery within three months
* Systemic disease
* Diagnosis of anemia

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of endogenous AAS metabolites | 1 week
  Doping substances in urine, mainly metabolites of anabolic androgenic steroids (AAS), were quantified, including testosterone (17β-hydroxyandrost-4-en-3-one), epitestosterone (17α- hydroxy-4-androsten-3-one), androsterone (4-androsten-3,17-dione), etiocholanolone (3α-hydroxy-5β-androstan-17-one), DHEA (dehydroepiandrosterone), dihydroandrosterone (5α- androstane-3α,17β-diol), and etiocholane-3α,17β-diol (5β -androstane-3α,17β-diol). Each urine sample (6 mL) was mixed with 50 μL standard solution and 1 mL phosphate buffer, and the mixture was heated for 60 min at 50°C. After cooling at room temperature, liquid-liquid extraction was performed, and phase separation was achieved. The organic extract was evaporated to dryness, and the dried residue was further derivatized with 50 μL of MSTFA solution for 30 min at 60°C. Finally, the sample was subjected to gas chromatographic analysis and mass spectrometric analysis for quantification of doping substances of interest.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Medical Hosptial, Kaohsiung City, Taiwan